CLINICAL TRIAL: NCT02924298
Title: Sit Less, Interact, Move More (SLIMM) Intervention Pilot Study
Brief Title: Effect of Sit Less, Interact, Move More (SLIMM) Regimen on Patients With Chronic Kidney Disease (CKD)
Acronym: SLIMM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Srinvasan Beddhu (Other)
Responsible Party: Sponsor-Investigator, Srinvasan Beddhu, MD, University of Utah
Organization: University of Utah (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00063835
Record Dates: First submitted 2014-01-06; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Kidney Disease; End Stage Renal Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stage 1-2 Chronic Kidney Disease (Experimental): Individuals with estimated glomerular filtration rate > 60 mL/min/1.73m^2, to undergo SLIMM intervention
  Interventions: Behavioral: SLIMM
- Stage 3-4 Chronic Kidney Disease (Experimental): Individuals with estimated glomerular filtration rate 15 to < 60 mL/min/1.73m^2, to undergo SLIMM intervention
  Interventions: Behavioral: SLIMM

INTERVENTIONS:
Behavioral: SLIMM — Participants will perform 5 minutes of light activity for every 25 minutes spent seated for 12 weeks. Following the week 12 visit, participants will increase light activity to 10 minutes for every 20 minutes spent seated.

SUMMARY:
In the past two decades, the prevalence of obesity in the US has increased from 23.2% to 32.9%. This epidemic is fueling the Chronic Kidney Disease (CKD) epidemic. This likely is the major challenge facing the nephrology community in the next decade and beyond. This pilot study is designed to test the feasibility of the Sit Less, Interact, Move More (SLIMM) intervention and to determine its preliminary impact on light physical activity (PA) levels. Increasing light PA may have significant impact on both obesity and slowing the progression of CDK.

DETAILED DESCRIPTION:
More than one-third of U.S. adults (35.7%) are obese (body mass index (BMI) > 30 kg/m2). In 2008, medical costs associated with obesity were estimated at $147 billion. Furthermore, there is a graded association of BMI and the risk of end stage renal disease (ESRD). Indeed, increasing prevalence of CKD in the US population is partly explained by increasing BMI. Hence, as a public health policy, it is imperative that obesity be targeted in order to decrease the morbidity, mortality and the healthcare costs burden associated with CKD and ESRD.

Physical inactivity plays a major role in obesity. Volitional exercise (VE), which includes moderate to vigorous physical activities (MVPA) such as sports and fitness-related activities, and non-volitional exercise, which includes low to light intensity physical activity (PA) such as activities of daily living, fidgeting, spontaneous muscle contraction, and maintaining posture in non-recumbent positions, represent two different ends of the PA spectrum. The current national recommendations are focused on MVPA (30 minutes of moderate PA five times a week or 25 minutes of vigorous activities three times a week). However, the relative importance of low and light activities and MVPA has not been established. As described in the preliminary data, the analyses of objectively measured PA in National Health And Nutrition Examination Survey (NHANES) suggest that a larger amount of light intensity PA is strongly associated with lower odds of proteinuria, lower odds of CKD and a lower hazard of death at any given level of MVPA. Furthermore, there appears to be a threshold effect for MVPA with mortality that plateaus at about half of the currently recommended levels of MVPA. Since physical function in the CKD population is low, 30 minutes of moderate PA five times a week or 25 minutes of vigorous activities three times a week might induce fatigue and paradoxically reduce light intensity PA. On the other hand, a lower target of MVPA might improve adherence with MVPA as well as not decrease light PA. This pilot intervention study will test the efficacy, feasibility and tolerability of the SLIMM intervention. The results of this intervention will be later used to determine if targeting obesity via the SLIMM intervention will slow kidney disease progression.

DESIGN:

This is a pilot intervention study that will examine the feasibility of and adherence to the SLIMM intervention to increase levels of light physical activity

Baseline visit: Baseline PA data will be collected by accelerometer in the week following the screening visit. Participants will be instructed on the importance of physical activity, the recommendations of 150 min/wk of moderate PA, or 75 min/wk of vigorous PA, and be provided with examples of physical activities.

SLIMM Intervention: The goal of the SLIMM intervention is to increase the time spent on light activities (Light physical activity is defined as 500-2019 counts/minute). This intervention will only be completed by individuals in the CKD and non-CKD groups. At week 6 of the intervention participants will be instructed to perform 5 minutes of light activity for each 25 minutes of sitting time. At week 12, participants will be instructed to further increase their light activity to a goal of 10 minutes for each 20 minute of sitting time. Thus, the goal is to replace total sedentary time by increase in light activities by 15% in 6 weeks and 33% by the end of the intervention.

All participants will undergo standardized training on the SLIMM intervention by trained study personnel at the 6 week visit. Participants will initially be asked to perform 5 minutes of light activity for every 25 minutes spent seated. At the week 12 visit, participants will be asked to further increase their activity, by performing 10 minutes of light activity for every 20 minutes spent seated.

Training will be provided in one to one sessions and reinforced at the following visits. Accelerometry data and paper PA diary data collected during the week before the baseline visit will be reviewed with the participant to provide feedback and used for devising a customized plan on increasing light activity. Examples of how to increase light activities within their natural, free-living environment will be provided. For instance, if the majority of their day is spent working at a desk, they will be encouraged to stand and/or walk for 5 minutes for every 25 minutes spent sedentary during weeks 6-12, and 10 minutes of light activity for every 20 minutes spent sedentary for weeks 12-18. Participants will be asked to stand and/or walk during commercial breaks when they are watching television.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be willing to participate in all study procedures and meet the criteria for one of the three groups listed below.

  1. Are currently receiving chronic maintenance dialysis
  2. Have CKD (eGFR 20 to 45 ml/min/1.73 m2 or eGFR > 45 and < 60 ml/min/1.73 m2)
  3. Individuals with eGFR >60 ml/min/1.73 m2

Exclusion Criteria:

* Age less than 18 years
* Pregnant women
* Prisoners
* Diagnosis of glomerulonephritis
* Life expectancy less than 1 year
* Expected to undergo renal replacement therapy within 1 year
* Enrolled in interventional trials using drugs or devices
* Physical mobility limitations that preclude physical activity interventions
* Individuals who are wheelchair bound, reliant on a walker or crutches for ambulation
* Patients who self-report MVOA greater than 150 min/week or more

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in level of light physical activity, measured in minutes per day | baseline to 18 weeks
  Determine the effect of SLIMM intervention as measured by the change in levels of light physical activity, measured by accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasan Beddhu, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Hsu CY, McCulloch CE, Iribarren C, Darbinian J, Go AS. Body mass index and risk for end-stage renal disease. Ann Intern Med. 2006 Jan 3;144(1):21-8. doi: 10.7326/0003-4819-144-1-200601030-00006. PMID 16389251
- [Background] Coresh J, Selvin E, Stevens LA, Manzi J, Kusek JW, Eggers P, Van Lente F, Levey AS. Prevalence of chronic kidney disease in the United States. JAMA. 2007 Nov 7;298(17):2038-47. doi: 10.1001/jama.298.17.2038. PMID 17986697
- [Background] Levine JA, Eberhardt NL, Jensen MD. Role of nonexercise activity thermogenesis in resistance to fat gain in humans. Science. 1999 Jan 8;283(5399):212-4. doi: 10.1126/science.283.5399.212. PMID 9880251
- [Background] Padilla J, Krasnoff J, Da Silva M, Hsu CY, Frassetto L, Johansen KL, Painter P. Physical functioning in patients with chronic kidney disease. J Nephrol. 2008 Jul-Aug;21(4):550-9. PMID 18651545
- [Background] Studenski S, Perera S, Wallace D, Chandler JM, Duncan PW, Rooney E, Fox M, Guralnik JM. Physical performance measures in the clinical setting. J Am Geriatr Soc. 2003 Mar;51(3):314-22. doi: 10.1046/j.1532-5415.2003.51104.x. PMID 12588574
- [Background] Tudor-Locke C, Ainsworth BE, Thompson RW, Matthews CE. Comparison of pedometer and accelerometer measures of free-living physical activity. Med Sci Sports Exerc. 2002 Dec;34(12):2045-51. doi: 10.1097/00005768-200212000-00027. PMID 12471314
- See also: Center for Disease Control and Prevention: Prevalence of Overweight, Obesity, and Extreme Obesity among Adults: United States Trends 1960-1962 through 2007-2008 — http://www.cdc.gov/nchs/data/hestat/obesity_adult_07_08/obesity_adult_07_08.pdf